CLINICAL TRIAL: NCT03567915
Title: Ultrasound Assessment of Gastric Emptying of Korean Meals in Healthy Volunteer: Rice and Noodle
Brief Title: Ultrasound Assessment of Gastric Emptying of Korean Meals: Rice and Noodle
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Dr, SMG-SNU Boramae Medical Center
Other Study IDs: 20180504
Record Dates: First submitted 2018-05-04; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Preoperative Fasting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rice: Group that healthy volunteers eat rice.
  Interventions: Other: Evaluation of gastric volume and content
- Noodle: Group that healthy volunteers eat noodle.
  Interventions: Other: Evaluation of gastric volume and content

INTERVENTIONS:
Other: Evaluation of gastric volume and content — The gastric volume and gastric content are assessed at 4, 5, 6, 7, and 8 hours after eating a meal.

SUMMARY:
The investigators evaluate gastric emptying time of common Korean meals (rice, noodles) in healthy volunteers.

DETAILED DESCRIPTION:
The investigators assess the gastric volume and contents of healthy volunteers at 4, 5, 6, 7, 8 hours after eating common Korean meal (rice or noodle) using a ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers

Exclusion Criteria:

* History of gastrectomy
* Anatomical abnormalities or mass of stomach

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-06-15 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Gastric emptying time | 1 hour
  The time for digesting a meal

SECONDARY OUTCOMES:
Incidence of full stomach | At 4, 5, 6, 7, and 8 hours after eating a meal.
  The incidence of full stomach is assessed by using ultrasonography.
Cross sectional area of the stomach | At 4, 5, 6, 7, and 8 hours after eating a meal.
  The cross sectional area of the stomach is assessed by using ultrasonography in the supine and right lateral positions.
Gastric volume | At 4, 5, 6, 7, and 8 hours after eating a meal.
  The volume of stomach is assessed using the following formula; volume of stomach (mL) = 27.0 + 14.6 x cross-sectional area (right lateral position) - 1.28 x age.
Type of gastric contents | At 4, 5, 6, 7, and 8 hours after eating a meal.
  The type of gastric contents is assessed using ultrasonography.